CLINICAL TRIAL: NCT05319288
Title: Treating Acute Low Back Pain With Acupuncture - Comparison of the Efficacy Between Distal Points and Local Points
Brief Title: Treating ALBP With Acupuncture - Comparison of the Efficacy Between Distal Points and Local Points
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hong Kong Baptist University (Other)
Responsible Party: Principal Investigator, Zhong Lidan, Assistant Professor, Hong Kong Baptist University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Acupuncture for ALBP
Record Dates: First submitted 2022-03-16; First posted 2022-04-08 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Low Back Pain
Keywords: Acute
MeSH Terms: conditions — Low Back Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Distal acupoints only group (Active Comparator): The DPOG (n=51) will receive acupuncture of distal acupoints only(SI3, EX-UE7) for ALBP.
  Interventions: Device: Acupuncture
- Local acupoints mainly combined with distal acupoints group (Active Comparator): LPMG (n=51) will receive acupuncture of local acupoints mainly(BL23, BL25, BL32) combined with distal points(BL40) for ALBP.
  Interventions: Device: Acupuncture

INTERVENTIONS:
Device: Acupuncture — In DPOG, motion style acupuncture would be used; in LPMG, Traditional Chinese Medicine acupuncture is used.

SUMMARY:
This study is a randomized controlled trial on acupuncture for Acute Low Back Pain(ALBP). According to literature, using distal acupoints only to treat ALBP is mostly recognized, but in our daily clinical practice, it is common to use local acupoints mainly combined with distal acupoints. Which method leads to better effect is one important clinical question in treating Low Back Pain(LBP) by acupuncture.

In this proposed study, the investigators aim to compare the efficacy of using "distal acupoints only" and "local acupoints mainly combined with distal acupoints" on ALBP.

DETAILED DESCRIPTION:
It will be a randomized controlled trial on acupuncture for ALBP, conducted at the Pok Oi Hospital - Hong Kong Baptist University Chinese Medicine Clinic cum Training and Research Centre (Kowloon City District) (KCDCMCTR). Registered Chinese Medicine Practitioner(RCMP) with at least two years of clinical experience and trained to treat participants in accordance with study protocols. 102 (18-65 years in age) participants with ALBP will be recruited from the public through advertisement and from the clinic (KCDCMCTR). Eligible participants will be randomly assigned to two groups. The participants are randomly allocated into two groups: distal acupoints only group(DPOG) and local acupoints mainly combined with distal acupoints group(LPMG). The DPOG (n=51) will receive acupuncture of distal acupoints only(SI3, EX-UE7). The LPMG (n=51) will receive acupuncture of local acupoints mainly(BL23, BL25, BL32) combined with distal points(BL40). Participants will be treated twice a week for a total of four weeks. Every participant will be administered 8 sessions of acupuncture. The primary outcome will be the change in low back pain intensity(in VAS scores) before and after the treatment. The secondary outcomes will be the Oswestry Disability Index. All outcomes will be evaluated at every session of treatment and the follow up period. Follow-up will be scheduled 1 month and 3 months after the completion of treatments. This clinical trial lasts 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Low Back Pain as chief complaint: pain and discomfort, localized below the costal margin and above the inferior gluteal folds, with or without leg pain;
* Participants' aged between 18 and 65 years old;
* Acute onset of symptom: lasting less than 6 weeks;
* Provided informed consent prior to the study.

Exclusion Criteria:

* Low back pain lasting more than 6 weeks;
* Alerting features (Red Flags) or serious conditions associated with acute low back pain: Significant trauma, unexplained weight loss, past history of malignancy, fever, age >65 years old, severe and unremitting night-time pain;
* Contraindication of acupuncture, including needle phobia, severe cutaneous condition, excessive hunger/exhaustion/overeat, emotional instability, pregnancy(relative contraindication) etc.;
* Received acupuncture treatment during the last month.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
low back pain intensity(in VAS scores) | before and four weeks after the treatment
  The primary outcome will be the change in low back pain intensity(in VAS scores) before and after the treatment.

SECONDARY OUTCOMES:
Oswestry Disability Index | before and four weeks after the treatment
  The secondary outcomes will be the Oswestry Disability Index.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhong Lidan, Kowloon Tong, Kowloon, Hong Kong